CLINICAL TRIAL: NCT07329634
Title: Randomized Evaluation of Neoadjuvant Stereotactic Radiosurgery (SRS) and Multi-fraction SRS Alone for the Treatment of Large Brain Metastases: A Polish Multicenter Trial Protocol
Brief Title: Evaluation of Neoadjuvant Stereotactic Radiosurgery (SRS) and Multi-fraction SRS Alone for the Treatment of Large Brain Metastases
Acronym: RENESANS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maciej Harat (Other)
Collaborators: Bydgoszcz University of Science and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Maciej Harat, Associate Professor of Radiation Oncology, Prof. Franciszek Lukaszczyk Memorial Oncology Center
Organization: Prof. Franciszek Lukaszczyk Memorial Oncology Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RENESANS01
Record Dates: First submitted 2025-09-02; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastasis
Keywords: Brain metastasis; Stereotactic radiosurgery; Neoadjuvant therapy; Multi-fraction therapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant SRS (Arm 1) (Experimental): Neoadjuvant SRS
  Interventions: Procedure: Neoadjuvant Stereotactic Body Radiation Therapy (SBRT)
- mfSRS alone (arm 2) (Active Comparator): mfSRS alone
  Interventions: Procedure: Multi-fraction Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Procedure: Neoadjuvant Stereotactic Body Radiation Therapy (SBRT) — Single dose of 12-16 Gy
  Arms: Neoadjuvant SRS (Arm 1)
Procedure: Multi-fraction Stereotactic Body Radiation Therapy (SBRT) — 30 Gy treatment in five fractions
  Arms: mfSRS alone (arm 2)

SUMMARY:
The prospective, two-arm, randomized, controlled, multicentric phase III RENESANS trial is designed to compare the efficacy and safety of neoadjuvant stereotactic radiosurgery (Neo-SRS) versus multi-fraction stereotactic radiosurgery (mfSRS) in patients with large brain metastases, with the primary objective of evaluating the incidence of central nervous system composite events.

DETAILED DESCRIPTION:
The RENESANS trial compares the efficacy and safety of two treatment strategies for large brain metastases: neoadjuvant stereotactic radiosurgery (Neo-SRS) and multi-fraction stereotactic radiosurgery (mfSRS) alone. It is a prospective, two-arm, randomized (1:1), controlled, multicentric phase III trial conducted between September 30, 2025 and September 30, 2033 in multiple radiation oncology units in Poland.

Study participants are patients with cancer and a Karnofsky performance status (KPS) >60 who have at least one brain metastasis appropriate for resection, not previously treated with SRS, and measuring ≥2.5 cm and <6 cm in the largest dimension. The intervention arms are: (i) neoadjuvant SRS (a single dose of 12-16 Gy SRS); and (ii) mfSRS alone (30 Gy delivered in 5 fractions).

The primary outcome is the number of participants developing a central nervous system (CNS) composite event, defined as local recurrence of the treated lesions, symptomatic radiation necrosis of the treated lesions, or development of leptomeningeal disease. Secondary outcomes include overall survival (OS), progression-free survival (PFS), adverse events assessed according to NCI CTCAE version 5.0 criteria, and health-related quality of life (QoL) assessed using the EORTC QLQ-C30 and QLQ-BN20 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* At least one brain metastasis appropriate for resection and not previously treated with SRS.
* Lesions ≥2.5 cm and ≤6 cm in largest dimension.
* Index lesion(s) will be treated, as outlined in the treatment section of the protocol.
* Seen by a neurosurgeon or radiation oncologist and judged to be appropriate for participation in this study, including the ability to tolerate Neo-SRS, i.e., the ability to lie flat in a stereotactic head mask.
* Any non-index lesion or lesions for which there is no possible resection must measure ≤4.0 cm in maximal dimension on the contrast MRI or CT brain scan obtained ≤35 days prior to pre-registration. Unresected lesions will be treated with SRS or mfSRS.
* KPS >60
* MRI confirms 1-10 lesions, one of which one is the index lesion. Each non-index lesion (up to nine) must measure ≤4 cm in maximal extent on contrast MRI and not otherwise require resection.
* Known active or history of invasive primary non-central nervous system (CNS) cancer based on a documented histopathological diagnosis within the past three years.
* Patient can tolerate surgery and SRS.
* History/physical examination within 14 days prior to registration.
* A negative urine or serum pregnancy test (in persons of childbearing potential, defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal for at least 12 consecutive months) within ≤14 days prior to registration.
* Participants who are sexually active must agree to use medically acceptable forms of contraception during treatment during this study to prevent pregnancy.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* No resectable lesion ≥2.5 cm.
* Unresectable >4 cm lesion.
* Previous whole brain irradiation.
* Progressive brain lesion treated with SRS.
* Previous resection of brain metastases.
* Leptomeningeal disease.
* Lesion diameter >6.0 cm, or more than 20 lesions in the brain.
* Required emergency decompressive surgery for life-threatening intracranial hypertension (with a preference towards adjuvant SRS/mfSRS protocols).
* Prior diagnosis of malignant brain tumor.
* Pediatric patients (age <18 years), pregnant women, and patients who are unable to give informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Central nervous system (CNS) composite event (CE) | From date of randomization to the date of a documented LR, SRN, or LMD, whichever comes first, assessed up to 12 months
  Number of participants experiencing a central nervous system (CNS) composite event (CE). A CNS CE is defined as the occurrence of at least one of the following events: local recurrence (LR) of a treated lesion, symptomatic radiation necrosis (SRN) of a treated lesion, or development of leptomeningeal disease (LMD). This is a composite endpoint analyzed as a single binary outcome per participant.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to the date of death or 12 months, whichever comes first
  OS is defined as the time between randomization and death due to any cause. Patients without an event will be censored at the date of last follow-up. Patients with no post-baseline follow-up for progression will be censored at the day of randomization. Median, six-month, and one-year OS will be measured
Progression-free survival (PFS) | From date of randomization to the date of death or 12 months, whichever comes first
  PFS is defined as the time from randomization until radiographic progression, based on Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria (including local recurrence and distant brain metastases), or death from any cause. Patients without an event will be censored at the date of last progression-free follow-up. Patients without post-baseline follow-up will be censored at the date of randomization. Median, 6-month, and 1-year PFS will be reported.
Incidence of adverse events (any grade) | From date of randomization to the date of death or 12 months, whichever occurs first
  All treatment-related adverse events (AEs) will be recorded from screening until disease progression or death. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. The number and proportion of participants experiencing at least one adverse event of any grade will be summarized by treatment arm.
Incidence of grade ≥3 adverse events | From date of randomization to the date of death or 12 months, whichever occurs first.
  The number and proportion of participants experiencing at least one treatment-related adverse event of grade 3 or higher, as defined by NCI CTCAE version 5.0, will be compared between treatment arms.
Health-related quality of life (EORTC QLQ-C30) | From date of randomization to the date of death or 12 months, whichever occurs first
  Health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Scores will be calculated according to the EORTC scoring manual and reported on a standardized scale from 0 to 100.
Brain-specific quality of life (EORTC QLQ-BN20) | From date of randomization to the date of death or 12 months, whichever occurs first.
  Brain cancer-specific quality of life will be assessed using the EORTC Brain Cancer Module (QLQ-BN20). Scores will be calculated according to the EORTC scoring manual and reported on a standardized scale from 0 to 100.

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication, no end date.
Access Criteria: Anyone who wishes to access the data.